CLINICAL TRIAL: NCT01146405
Title: Memory During Anesthesia: the Role of Stress Hormones
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Liliana Sollazzi, Catholic University of Sacred Heart
Other Study IDs: 918/09
Record Dates: First submitted 2010-06-09; First posted 2010-06-17 (Estimated); Last update posted 2011-02-09 (Estimated); Status verified 2009-10

CONDITIONS: Surgical Procedure, Unspecified
Keywords: Laparoscopic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood and serum.
Oversight: Data Monitoring Committee: No

SUMMARY:
1. To investigate whether the auditory stimulation causes changes in hormones levels (cortisol+prolactin) during general anesthesia.
2. To determine if there is a correlation between hormones levels (cortisol+prolactin) and dreams recall.
3. To investigate whether, in patients receiving auditory stimulation, there is a correlation between hormones levels (cortisol+prolactin), serum remifentanil concentration and detection of implicit memory.
4. To investigate the presence of primary auditory cortex activation (temporal lobe) in patients with implicit memory and in those with dreams recall using the EEG-ERP 128 channels GES300 EGI system.

DETAILED DESCRIPTION:
Patients from group A, during maintenance of anesthesia, at the time of trocar insertion, will listen (via MP3) a piece of one of two stories, "Puss in Boots" and "Pinocchio", each followed by four keywords. In group B, patients will be isolated from the sounds of the operating room using specific headphones.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years old
* Class-ASA Physical Status I-II

Exclusion Criteria:

* Psychiatric or neurological disorders and/or hearing disorders
* Obesity (Body Mass Index > 30)
* Drug addiction, alcoholism
* Patients with an education level below middle school
* Patients with difficulty in understanding the Italian language
* Patients treated with corticosteroids and/or estrogens, pregnant patients and patients suffering from hypercorticism

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients sheduled for minor elective laparoscopic surgery
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-10 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Hormones levels | 5 minutes after achieving a pneumoperitoneum pressure of 12 mmHg
  The blood sample will be taken during anaesthesia to determine intraoperative hormones (cortisol + prolactine) levels.
Hormones levels | Baseline
  The blood sample will be taken 30 minutes before induction of anaesthesia to determine baseline hormones (cortisol + prolactine) levels.

SECONDARY OUTCOMES:
Remifentanil concentration | 5 minutes after achieving a pneumoperitoneum pressure of 12 mmHg
  One blood sample will be taken to determine steady state concentration of remifentanil (only in a subset of patients).
Memory | Approximately 24 hours after surgery for explicit memory, implicit memory and for dreams recall detected after awakening from anesthesia
  Patients will be asked to associate with keywords the first thing that comes them to mind (implicit memory). Also eplicit memory and dreams recall will be tested at the same time. The content of intraoperative dreams (confirmed by a brief post-anesthesia interview) will be analyzed using the 5-point Likert scale.
Primary auditory cortex activation | 5 minutes after achieving a pneumoperitoneum pressure of 12 mmHg
  ERP-EEG monitoring system with 128 channel EGI GES300

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Sacred Heart, Rome, Italy